CLINICAL TRIAL: NCT06235593
Title: Self-care in the Person With Chronic Disease: A Protocol for a Self-care Intervention
Brief Title: Self-care in the Person With Chronic Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Cláudia Mendes, Principal Investigator, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRC052023
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Disease; Self-Control
Keywords: Illness, Chronic; quality of life; elderly
MeSH Terms: conditions — Chronic Disease; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The intervention will be a combination of interviews and face-to-face follow-ups, with teleconsultations, based on other observational and experimental studies. The intervention program includes monitoring for 9 months
  Interventions: Behavioral: Self-care Intervention

INTERVENTIONS:
Behavioral: Self-care Intervention — The intervention will focus on self-care behavior of people with chronic diseases according to two distinct periods (through a longitudinal study - follow-up nursing interventions):
  (i) baseline; and (ii) 4 months;

SUMMARY:
Determine the nursing care needs of the elderly population sample according to the self-care deficits identified using the "Self-Care of Chronic Illness Inventory - Patient Version (version 4)" in elderly population living in their own homes or in the homes of relatives or friends in the district of Évora.

DETAILED DESCRIPTION:
An assessment of the Portuguese health system estimates the overall burden of chronic diseases in the Portuguese population (regardless of age/gender) is follows: (i) 18% of Portuguese users of the National Health System have one chronic disease, (ii) 11% of users have two chronic diseases, (iii) 8% of users have three chronic diseases, and (iv) 22% of users have four or more chronic diseases; therefore, at least 59% of the Portuguese population has one or more chronic diseases (estimate). Moreover, the same report reveals that multimorbidity increases with age, with a maximum between 80 and 90 years old. Moreover, according to the research published in 2019 concerning the first National Health Examination Survey, the authors reported a high prevalence of multimorbidity among individuals aged 65 and older, estimated at 78.3% for the Portuguese population sample used in their research (estimates reported by age groups of 65-69, 70-74, 75-79 and 80 years and older: 72.8%, 78.2%, 81.9%, and 83.4%, respectively). Studying individual aging by integrating a continuous and accessible care model that allows elderly individuals as well as family caregivers to monitor and manage their health at home- always under the supervision of health professionals, which may enable the management of various chronic conditions (multimorbidity) and provide a "safety net" before a health crisis requiring emergency department care occurs. To promote improved health-related quality of life among elderly individuals by requalifying their potential and allowing them to live more autonomously, the following tasks are essential to identify the appropriate self-care behavior that allows determining, planning, and assessing preventive nursing care needs. Health care for patients with multimorbidity and applicable intervention strategies yield better outcomes when structured based on a previous evaluation of the patient's self-care deficits.

Most aging populations report chronic illnesses, which are usually permanent or recurrent, significantly affect well-being and quality of life, require daily and consistent healthcare management and last more than three months. With chronic illness now the significant health threat and the primary driver of healthcare costs, researchers, healthcare providers, and payers are focusing on interventions that can prevent or control exacerbations. In this context, the importance of self-care is increasingly recognized.

Self-care is essential in aging, mainly when changes occur in the person's health condition. Theoretically, this process involves three linked sequential behaviors captured in the critical concepts of self-care maintenance, self-care monitoring, and self-care management. Self-care maintenance addresses behaviors used by patients with a chronic illness to maintain physical and emotional stability (e.g., medication adherence), while self-care monitoring involves the behavior of observing oneself for signs and symptoms(e.g., checking blood pressure). Self-care monitoring is the link or bridge between self-care maintenance and self-care management. A core goal of self-care monitoring is symptom recognition; once recognized, self-care management (e.g., taking medicine for a symptom) can occur, with behaviors that reflect a response to the observed symptoms. There are two approaches to measurement: generic and disease-specific. Generic measures apply to a wide variety of patients. Disease-specific measures are helpful in specific groups with a single condition. Disease-specific measures are more responsive because they target issues experienced by patients with an explicit condition. Generic measures allow comparison among patients with different conditions and accommodate those with more than one diagnosis. The instrument studied within this project's scope, the "Self-Care of Chronic Illness Inventory - Patient Version" (version 4), is a generic measure designed to assess the process of self-care used by individuals with various chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* are aged 65 or older
* are interested in participating in the project
* are residing Évora district in their own homes or at family members' or friends' homes
* can make their own decisions if they were sick or were hospitalized due to acute, short-term health care needs
* present at least one chronic disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Self-Care Maintenance | 9 months
  Eigth items questionnaire - Self-Care of Chronic Illness Inventory - Patient Version; Minimum -1 value and maximum- 5 value; higher scores mean a better outcomes.
Self-Care Monitoring | 9 months
  Six items questionnaire - Self-Care of Chronic Illness Inventory - Patient Version; Minimum -1 value and maximum- 5 value; higher scores mean a better outcomes.
Self-Care Management | 9 months
  Six items questionnaire - Self-Care of Chronic Illness Inventory - Patient Version; Minimum -1 value and maximum- 5 value; higher scores mean a better outcomes.

SECONDARY OUTCOMES:
Health-related Quality of life | 9 months
  Quality of life will be assessed using the WHOQOL-BREF(PT); Minimum - 0 value and maximum- 100 value; higher scores mean a better outcomes.
  Quality of life will be assessed using the general health and well-being questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
The group plans to share all data after the individual project validation

REFERENCES:
- [Result] Quinaz Romana G, Kislaya I, Salvador MR, Cunha Goncalves S, Nunes B, Dias C. [Multimorbidity in Portugal: Results from The First National Health Examination Survey]. Acta Med Port. 2019 Feb 1;32(1):30-37. doi: 10.20344/amp.11227. Epub 2019 Feb 1. Portuguese. PMID 30753801
- [Result] Gruneir A, Silver MJ, Rochon PA. Emergency department use by older adults: a literature review on trends, appropriateness, and consequences of unmet health care needs. Med Care Res Rev. 2011 Apr;68(2):131-55. doi: 10.1177/1077558710379422. Epub 2010 Sep 9. PMID 20829235
- [Result] Goes M, Lopes MJ, Oliveira H, Fonseca C, Maroco J. A Nursing Care Intervention Model for Elderly People to Ascertain General Profiles of Functionality and Self Care Needs. Sci Rep. 2020 Feb 4;10(1):1770. doi: 10.1038/s41598-020-58596-1. PMID 32019984
- [Result] Martin Lesende I, Mendibil Crespo LI, Castano Manzanares S, Otter AD, Garaizar Bilbao I, Pison Rodriguez J, Negrete Perez I, Sarduy Azcoaga I, de la Rua Fernandez MJ. Functional decline and associated factors in patients with multimorbidity at 8 months of follow-up in primary care: the functionality in pluripathological patients (FUNCIPLUR) longitudinal descriptive study. BMJ Open. 2018 Jul 28;8(7):e022377. doi: 10.1136/bmjopen-2018-022377. PMID 30056392
- [Result] Goes M, Lopes M, Maroco J, Oliveira H, Fonseca C. Psychometric properties of the WHOQOL-BREF(PT) in a sample of elderly citizens. Health Qual Life Outcomes. 2021 May 17;19(1):146. doi: 10.1186/s12955-021-01783-z. PMID 34001152
- [Result] Luciani M, De Maria M, Page SD, Barbaranelli C, Ausili D, Riegel B. Measuring self-care in the general adult population: development and psychometric testing of the Self-Care Inventory. BMC Public Health. 2022 Mar 28;22(1):598. doi: 10.1186/s12889-022-12913-7. PMID 35346104
- [Result] Riegel B, De Maria M, Barbaranelli C, Matarese M, Ausili D, Stromberg A, Vellone E, Jaarsma T. Symptom Recognition as a Mediator in the Self-Care of Chronic Illness. Front Public Health. 2022 May 17;10:883299. doi: 10.3389/fpubh.2022.883299. eCollection 2022. PMID 35655456
- [Result] Okubo K, Sei Y, Matsuo Y, Sagawa K, Natori H, Yokoyama MM. [Tac antigen expression on non-T non-B acute lymphocytic leukemia cells]. Nihon Ketsueki Gakkai Zasshi. 1985 May;48(3):794-801. No abstract available. Japanese. PMID 2994340
- [Result] Porter ME, Larsson S, Lee TH. Standardizing Patient Outcomes Measurement. N Engl J Med. 2016 Feb 11;374(6):504-6. doi: 10.1056/NEJMp1511701. No abstract available. PMID 26863351